CLINICAL TRIAL: NCT07137013
Title: Evaluation of the Relationship Between Periodontal Disease Severity and Retinal Layer Thickness in Patients With Diabetic Retinopathy Using Optical Coherence Tomography
Brief Title: Periodontitis Severity in Patients With Diabetic Retinopathy
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Dilek KARADOĞAN, Assoc. Prof. Dr., Recep Tayyip Erdogan University Training and Research Hospital
Other Study IDs: DR2025/59
Record Dates: First submitted 2025-08-11; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Diabetic Retinopathy; Periodontitis
Keywords: Diabetic Retinopathy; Periodontitis; Optical Coherence Tomography; Optical Coherence Tomography Angiography
MeSH Terms: conditions — Diabetic Retinopathy; Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Control: without systemic disease
- DM+ DR-: Diagnosed with Diabetes Mellitus and not diagnosed with Diabetic Retinopathy
- NPDR+ DMÖ-: Diagnosed with non-proliferative Diabetic Retinopathy without diabetic macular edema
- NPDR+ DMÖ+: Diagnosed with non-proliferative DR with diabetic macular edema
- PDR: Diagnosed with proliferative Diabetic Retinopathy

SUMMARY:
The aim of this observational study is to investigate the relationship between periodontal disease severity and retinal layer thickness in patients diagnosed with diabetic retinopathy (DR), using optical coherence tomography (OCT) for assessment.

The main question this study seeks to answer is:

Do measurable changes in retinal layer thickness occur as periodontal disease severity increases in patients with diabetic retinopathy?

Participants will include adult individuals with a confirmed clinical diagnosis of DR. Periodontal status will be assessed through standard clinical parameters, including plaque index, probing pocket depth, clinical attachment loss, and bleeding on probing. Retinal layer thickness will be measured using high-resolution OCT and OCT angiography (OCTA) devices. The study aims to analyze potential associations between periodontal disease severity and morphological as well as vascular changes in the retina.

DETAILED DESCRIPTION:
This observational study will aim to evaluate the possible relationship between periodontal disease severity and retinal layer thickness in patients with diabetic retinopathy (DR). Adult individuals with a confirmed clinical diagnosis of DR will be included in the study. Periodontal health status will be assessed using standard clinical parameters such as plaque index, probing pocket depth, clinical attachment loss, and bleeding on probing. Retinal layer thickness will be measured using high-resolution imaging with optical coherence tomography (OCT). Optical coherence tomography angiography (OCTA) will be used to evaluate vascular changes. The collected data will be analyzed to determine whether periodontal disease severity is associated with possible changes in retinal morphology and vascularity. This study is expected to provide new scientific evidence on the interaction between systemic diabetic complications and oral health, as well as to highlight the importance of multidisciplinary approaches.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 and over
* Those without systemic disease (control group)
* Patients diagnosed with diabetic retinopathy
* Patients diagnosed with diabetes mellitus (HbA1c>6)

Exclusion Criteria:

* Patients with any autoimmune disease, osteoporosis, or cancer
* Patients taking immunosuppressive medications, oral contraceptives, or bisphosphonates
* Pregnancy
* Patients with acute or chronic eye diseases such as vitreoretinal, optic nerve, or choroidal vascular diseases, cataracts, glaucoma, retinal degeneration, uveitis, Behçet's disease, or scleritis
* Patients undergoing refractive or intraocular surgery
* Presence of active infectious disease (acute hepatitis, tuberculosis, AIDS)
* Chronic use of medications affecting periodontal tissues (cyclosporine A, phenytoin)
* Patients taking antioxidant supplements

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals over the age of 60 who apply to the Department of Ophthalmology at Recep Tayyip Erdoğan University Faculty of Medicine
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Optical Coherence Tomography (OCT) Measurement | Day 1
  A macular thickness map (ETDRS = Early Treatment Diabetic Retinopathy Study) is examined using OCT, with the center at the fovea centralis. According to the ETDRS map, the central 1 mm represents the fovea, the surrounding 3 mm area represents the inner retinal layers, and the outermost 6 mm area represents the outer retinal layers.
Optical Coherence Tomography Angiography (OCTA) Measurement | Day 1
  OCTA is a non-invasive technique that allows the evaluation of microvascular changes at the capillary level and imaging of the retinal plexuses layer by layer.
Retinal Layer Thickness | Day 1
  Definition: Retinal thickness is the distance between the internal limiting membrane (ILM) and the retinal pigment epithelium (RPE), measured by optical coherence tomography (OCT).
  ETDRS Mapping: The macular region is divided into nine sectors based on the ETDRS grid:
  Central subfield: A 1 mm diameter circle centered on the fovea. Inner ring (parafoveal region): 1-3 mm diameter, divided into superior, inferior, nasal, and temporal quadrants.
  Outer ring (perifoveal region): 3-6 mm diameter, also divided into four quadrants.
Choroidal Thickness (CSI Reference) | Day 1
  Definition: The choroid is the vascular layer beneath the RPE. Choroidal thickness is the perpendicular distance from Bruch's membrane to the choroid-sclera interface (CSI).
  Measurement: Typically obtained with enhanced depth imaging OCT (EDI-OCT), mapped according to the ETDRS grid.
Ganglion Cell Layer (GCL) Thickness | Day 1
  Definition: The GCL is composed of the cell bodies of retinal ganglion cells, located between the inner plexiform layer and the retinal nerve fiber layer.
  Measurement: OCT can quantify GCL alone or GCL + inner plexiform layer (GCL+IPL), usually reported using the ETDRS 9-sector mapping.
Retinal Nerve Fiber Layer (RNFL) Thickness | Day 1
  Definition: The RNFL consists of the unmyelinated axons of ganglion cells, located at the innermost surface of the retina.
  Measurement: Often assessed in the peripapillary region or in the macular area using ETDRS mapping.
Choroid-Sclera Interface (CSI) | Day 1
  Definition: The CSI is the outer anatomical boundary of the choroid where it transitions into the sclera.
  Role in Thickness Measurement: Serves as the lower reference point for choroidal thickness measurements (Bruch's membrane to CSI), which can be mapped according to the ETDRS grid.
Superficial Retinal Layers | Day 1
  Definition: The inner portion of the retina, located closer to the vitreous side.
  Typically associated with the superficial capillary plexus. These layers are among the first affected in diseases such as glaucoma, optic neuropathies, and ischemic retinopathies.
Deep Retinal Layers | Day 1
  Definition: The middle and outer portions of the retina, located closer to the photoreceptors.
  Associated with the deep capillary plexus. Clinical relevance: Important changes are observed here in conditions such as macular edema, diabetic retinopathy, and age-related macular degeneration.
Foveal Avascular Zone (FAZ) | Day 1
  Definition: A circular area at the center of the fovea devoid of retinal capillary vessels.
  Location: In the central fovea, approximately 500-600 micrometers in diameter.
  Characteristics:
  Contains the highest density of photoreceptors (especially cones). Avascular nature means nutrition is supplied via diffusion from the choroid. Responsible for the highest visual acuity. Clinical relevance: FAZ size, measurable by OCT angiography (OCTA), is an important biomarker in diabetic retinopathy, retinal vein occlusion, and macular ischemia.

SECONDARY OUTCOMES:
Clinical Periodontal Parameters (Plaque Index) | Day 1
  Plaque Index (PI) (Silness and Löe, 1964) This index is used to evaluate the amount of dental plaque accumulation on tooth surfaces. Each tooth's four surfaces (buccal, lingual, mesial, distal) are examined using a probe or visually. Each surface is scored from 0 to 3. The average score is calculated for each tooth. The overall plaque index is obtained by averaging the scores from all examined teeth.
  Score Description 0 No plaque.
  1. No visible plaque, but a slight film of plaque is detected when a probe is run along the gingival margin.
  2. Visible plaque along the gingival margin, forming a continuous band.
  3. Abundant plaque covering the gingival area and extending toward the middle of the tooth surface, including the interproximal spaces.
Clinical Periodontal Parameters (Gingival Index) | Day 1
  The Gingival Index is used to assess the presence and severity of gingival inflammation (gingivitis). Four surfaces of each tooth (buccal, lingual, mesial, distal) are examined visually and with a periodontal probe. The evaluation considers color changes, edema (swelling), tissue consistency, and bleeding on probing. Each surface is scored from 0 to 3. The average score per tooth is calculated, and then the overall average is used to determine the individual's GI score.
  Score Description 0 Healthy gingiva: normal color and texture, no bleeding
  1. Mild inflammation: slight color change and swelling, no bleeding on probing
  2. Moderate inflammation: redness, edema, soft tissue, bleeding on probing
  3. Severe inflammation: marked redness and swelling, ulceration, possible spontaneous bleeding
Periodontal Clinical Parametres (Bleeding on Probing Index) | Day 1
  This index is used to assess the presence and severity of gingival inflammation by observing bleeding after gentle pressure is applied to the gingival sulcus using a periodontal probe. A thin periodontal probe is gently inserted into the gingival sulcus with light pressure (approximately 20-25 grams). Bleeding occurring within 10-30 seconds is observed. Each measurement site is recorded as either "bleeding present" or "bleeding absent." Presence of bleeding is an early and sensitive indicator of gingival inflammation.
  Score Description: 0 No bleeding 1 Bleeding present (mild or severe)
Periodontal Clinical Parametres (Probing Pocket Depth) | Day 1
  Using a Williams periodontal probe, the distance between the gingival margin and the base of the periodontal pocket is measured in millimeters at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual. All teeth are measured. The values obtained from each site are summed and then divided by the total number of sites measured. This gives the average probing depth for the individual.
  Measurement Interpretation 1-3 mm Healthy sulcus 4-5 mm Shallow to moderate pocket
  ≥6 mm Deep periodontal pocket (advanced disease)
Periodontal Clinical Parametres (Clinical Attachment Loss) | Day 1
  Using a Williams periodontal probe, the distance between the enamel-cementum junction and the base of the periodontal pocket is measured in millimeters at six sites per tooth: mesiobuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual. All teeth are measured. The values obtained from each site are summed and then divided by the total number of sites measured. This gives the average probing depth for the individual.
  CAL Value Interpretation 0-1 mm Healthy / minimal loss 2-3 mm Mild attachment loss 4-5 mm Moderate attachment loss
  ≥6 mm Severe attachment loss

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology of the Faculty of Medicine of Recep Tayyip Erdogan University, Rize, Rize Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No